CLINICAL TRIAL: NCT02910050
Title: A Phase II Study of the Efficacy and Tolerability of Bicalutamide Plus Aromatase Inhibitors in Estrogen Receptor(+)/Androgen Receptor(+)/HER2(-) Metastatic Breast Cancer
Brief Title: Bicalutamide Plus Aromatase Inhibitors in ER(+)/AR(+)/HER2(-) Metastatic Breast Cancer
Acronym: BETTER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu fei (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Xu fei, associate chief physician,associate professor,MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU5010-2016
Record Dates: First submitted 2016-09-06; First posted 2016-09-21 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: androgen receptor; bicalutamide; aromatase inhibitors; advanced breast cancer; letrozole; anastrozole; exemestane
MeSH Terms: conditions — Breast Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — bicalutamide; Aromatase Inhibitors; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bicalutamide+ Aromatase Inhibitor (Experimental): ER(+)/AR(+)/HER2(+) metastatic breast cancer patients that previously treated by an aromatase inhibitor
  Interventions: Drug: Bicalutamide; Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Bicalutamide — 50mg once a day orally
  Other Names: Casodex
Drug: Aromatase Inhibitor — participants will receive any kind of aromatase inhibitor which has not been received before (steroidal AI change to nonsteroidal AI and vice versa), Letrozole 2.5mg once a day orally, Anastrozole 1mg once a day orally, Exemestane 25mg once a day orally
  Other Names: letrozole; anastrozole; exemestane

SUMMARY:
This study is aim to evaluate the efficacy and safety of bicalutamide and aromatase inhibitor in ER(+)/AR(+)/HER2(-) metastatic breast cancer patients who have disease progression after treatment of an aromatase inhibitor.

DETAILED DESCRIPTION:
Androgen receptor(AR) is closely related to molecular type, treatment and prognosis in breast cancer. Over 70% of breast cancer expressed androgen receptor. And in some estrogen receptor positive breast cancer cells which are resistant to Aromatase inhibitors can change androgen receptor dependent. So AR may be a new target in the treatment of breast cancer. Bicalutamide is a selective androgen receptor inhibitor with a clinical benefit rate of 19% and median progression free survival of 12 weeks in the ER-/AR+ metastatic breast cancer. This study is aim to evaluate the efficacy and safety of bicalutamide and aromatase inhibitor in ER+/AR+/HER- metastatic breast cancer patients who have disease progression after treatment of an AI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed estrogen receptor positive, androgen positive and HER2 negative breast cancer
* Metastatic or unresectable locally advanced disease
* Age over 18 years
* Postmenopausal status （continuous using luteinizing hormone releasing hormone(LHRH) analogue is available）
* Patient must have disease progression after treatment of an Aromatase inhibitor.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS)0-2
* Life expectancy over 3 months.
* Measurable disease according to RECIST version 1.1 or only bone metastasis
* Adequate hematological, hepatic function.
* Voluntarily signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

* Patient with life-threatening visceral metastasis, such as extensive liver metastasis, brain or meningeal metastasis
* Concomitant diseases/conditions that is not controllable, and Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
* History of other primary malignancy
* Resistant to steroidal or nonsteroidal aromatase Inhibitor

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
clinical benefit rate（CBR） | 24 weeks
  Response and progression will be evaluated using RECIST 1.1. Evaluation will occur every 2 months for the first 6 months and then every 3 months till progression or termination of the study.CBR is defined as ratio of participants who have stable disease for over 24 weeks.

SECONDARY OUTCOMES:
progression free survival | baseline up to approximately 6 months
  Time from to the first documentation of objective tumor progression or to death due to any cause.
objective response rate of bicalutamide plus another AI in participants with measurable disease | 24 weeks
  objective response rate includes complete response, partial response.
tolerability of bicalutamide plus an Aromatase inhibitor | 2 years
  evaluate and quality of life of the participants using Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) .

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- State Key Laboratory of Oncology in South China,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuenen-Boumeester V, Van der Kwast TH, Claassen CC, Look MP, Liem GS, Klijn JG, Henzen-Logmans SC. The clinical significance of androgen receptors in breast cancer and their relation to histological and cell biological parameters. Eur J Cancer. 1996 Aug;32A(9):1560-5. doi: 10.1016/0959-8049(96)00112-8. PMID 8911118
- [Background] Mangelsdorf DJ, Thummel C, Beato M, Herrlich P, Schutz G, Umesono K, Blumberg B, Kastner P, Mark M, Chambon P, Evans RM. The nuclear receptor superfamily: the second decade. Cell. 1995 Dec 15;83(6):835-9. doi: 10.1016/0092-8674(95)90199-x. No abstract available. PMID 8521507
- [Background] Grogg A, Trippel M, Pfaltz K, Ladrach C, Droeser RA, Cihoric N, Salhia B, Zweifel M, Tapia C. Androgen receptor status is highly conserved during tumor progression of breast cancer. BMC Cancer. 2015 Nov 9;15:872. doi: 10.1186/s12885-015-1897-2. PMID 26552477
- [Background] Brys M. Androgens and androgen receptor: do they play a role in breast cancer? Med Sci Monit. 2000 Mar-Apr;6(2):433-8. PMID 11208351
- [Background] Witzel I, Graeser M, Karn T, Schmidt M, Wirtz R, Schutze D, Rausch A, Janicke F, Milde-Langosch K, Muller V. Androgen receptor expression is a predictive marker in chemotherapy-treated patients with endocrine receptor-positive primary breast cancers. J Cancer Res Clin Oncol. 2013 May;139(5):809-16. doi: 10.1007/s00432-013-1382-8. Epub 2013 Feb 8. PMID 23392859
- [Background] Fujii R, Hanamura T, Suzuki T, Gohno T, Shibahara Y, Niwa T, Yamaguchi Y, Ohnuki K, Kakugawa Y, Hirakawa H, Ishida T, Sasano H, Ohuchi N, Hayashi S. Increased androgen receptor activity and cell proliferation in aromatase inhibitor-resistant breast carcinoma. J Steroid Biochem Mol Biol. 2014 Oct;144 Pt B:513-22. doi: 10.1016/j.jsbmb.2014.08.019. Epub 2014 Aug 29. PMID 25178713
- [Background] Ciupek A, Rechoum Y, Gu G, Gelsomino L, Beyer AR, Brusco L, Covington KR, Tsimelzon A, Fuqua SA. Androgen receptor promotes tamoxifen agonist activity by activation of EGFR in ERalpha-positive breast cancer. Breast Cancer Res Treat. 2015 Nov;154(2):225-37. doi: 10.1007/s10549-015-3609-7. Epub 2015 Oct 20. PMID 26487496
- [Background] Cuenca-Lopez MD, Montero JC, Morales JC, Prat A, Pandiella A, Ocana A. Phospho-kinase profile of triple negative breast cancer and androgen receptor signaling. BMC Cancer. 2014 Apr 30;14:302. doi: 10.1186/1471-2407-14-302. PMID 24779793
- [Background] Garay JP, Karakas B, Abukhdeir AM, Cosgrove DP, Gustin JP, Higgins MJ, Konishi H, Konishi Y, Lauring J, Mohseni M, Wang GM, Jelovac D, Weeraratna A, Sherman Baust CA, Morin PJ, Toubaji A, Meeker A, De Marzo AM, Lewis G, Subhawong A, Argani P, Park BH. The growth response to androgen receptor signaling in ERalpha-negative human breast cells is dependent on p21 and mediated by MAPK activation. Breast Cancer Res. 2012 Feb 9;14(1):R27. doi: 10.1186/bcr3112. PMID 22321971
- [Background] Tarulli GA, Butler LM, Tilley WD, Hickey TE. Bringing androgens up a NOTCH in breast cancer. Endocr Relat Cancer. 2014 Aug;21(4):T183-202. doi: 10.1530/ERC-14-0248. Epub 2014 Jul 7. PMID 25001242
- [Background] Ueda T, Bruchovsky N, Sadar MD. Activation of the androgen receptor N-terminal domain by interleukin-6 via MAPK and STAT3 signal transduction pathways. J Biol Chem. 2002 Mar 1;277(9):7076-85. doi: 10.1074/jbc.M108255200. Epub 2001 Dec 19. PMID 11751884
- [Background] Gucalp A, Tolaney S, Isakoff SJ, Ingle JN, Liu MC, Carey LA, Blackwell K, Rugo H, Nabell L, Forero A, Stearns V, Doane AS, Danso M, Moynahan ME, Momen LF, Gonzalez JM, Akhtar A, Giri DD, Patil S, Feigin KN, Hudis CA, Traina TA; Translational Breast Cancer Research Consortium (TBCRC 011). Phase II trial of bicalutamide in patients with androgen receptor-positive, estrogen receptor-negative metastatic Breast Cancer. Clin Cancer Res. 2013 Oct 1;19(19):5505-12. doi: 10.1158/1078-0432.CCR-12-3327. Epub 2013 Aug 21. PMID 23965901
- [Derived] Lu Q, Xia W, Lee K, Zhang J, Yuan H, Yuan Z, Shi Y, Wang S, Xu F. Bicalutamide plus Aromatase Inhibitor in Patients with Estrogen Receptor-Positive/Androgen Receptor-Positive Advanced Breast Cancer. Oncologist. 2020 Jan;25(1):21-e15. doi: 10.1634/theoncologist.2019-0564. Epub 2019 Aug 21. PMID 31434793